CLINICAL TRIAL: NCT06125392
Title: A Multicenter RegIstry on the Diagnosis of Patients with Chronic Angina and No Angiographic CoRonary Artery Stenosis (international Retrospective Collection of Anonymized Patient Data) - Searching a New Ach Spasm Definition
Brief Title: Multicenter Registry on Microvascular Dysfunction - Searching a New Ach Spasm Definition
Acronym: MICRO-SNAPE
Status: Recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Professor, Johannes Gutenberg University Mainz
Other Study IDs: UM 20-0274
Record Dates: First submitted 2023-09-26; First posted 2023-11-09 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Coronary Microvascular Disease; Coronary Vasospasm
MeSH Terms: conditions — Microvascular Angina; Coronary Vasospasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Invasive assessment of coronary vasomotor function: All lesions undergoing assessment of coronary microvascular dysfunction and coronary spasm using coronary pressure wires.
  Interventions: Diagnostic Test: Coronary physiology assessment

INTERVENTIONS:
Diagnostic Test: Coronary physiology assessment — Resting distal coronary to aortic pressure ratio, resting flow ratio, fractional flow reserve, Coronary Flow Reserve and Microvascular resistance using the thermodilution method and papaverin or adenosine, Resting distal coronary to aortic pressure ratio, resting flow ratio, fractional flow reserve, Coronary Flow Reserve and Microvascular resistance using the thermodilution method and acetylcholine.
  Other Names: Parameters of coronary physiology in response to microvascular vasodilators (adenosine, papaverine) and acetylcholine

SUMMARY:
The MICRO-SNAPE registry will collect data from patients undergoing investigation of microvascular dysfunction and coronary spasm in Europe and North America.

DETAILED DESCRIPTION:
Microvascular dysfunction is an important determinant of patients´quality of life and prognosis, which however remains poorly classified. Given the high burden of disease and the severity of the functional impairment in these patients, the lack of a clear understanding and diagnosis has a potentially large clinical importance. It is therefore important to better describe the phenotype of these patients. The MICRO-SNAPE registry will allow investigating these associations. Patient data as collected during the local clinical practice and at the operator's discretion, will be retrospectively entered in this non-interventional registry in anonymous form.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent combined measurements of coronary pressure and flow in at least 1 native coronary artery in response to endothelium dependent and independent vasodilators.

Exclusion Criteria:

* Hemodynamic instability
* Age <18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angina but no epicardial disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Identification of endotypes of coronary vasomotor function | immediately after the invasive measurement
  Patients will be classified in different endotypes according to the pattern of their responses to endothelium-dependent and independent vasodilators.

SECONDARY OUTCOMES:
Accuracy of clinical criteria for the diagnosis of microvascular and epicardial spasm | immediately after the invasive measurement
  The clinical criteria commonly used for the diagnosis of spasm (based on ECG and angina) will be validated against the benchmark invasive measurements
Normal values expressing endothelium-dependent coronary flow reserve | immediately after the invasive measurement
  Acetylcholine-induced coronary flow reserve in subjects without microvascular dysfunction.
Sex impact on coronary vasospasm measures | immediately after the invasive measurement
  Difference between males and females in microvascular and epicardial spasm measures
Coronary bridge and epicardial spasm | immediately after the invasive measurement
  Impact of coronary brudge on the incidence of epicaridal spasm
Acetylcholine versus adenosine responses | immediately after the invasive measurement
  Comparison of adenosine- versus acetylcholin-induced microvascular dilatation (IMR)
Normal values and associations of resting microvascular resistances | Immediately upon measurment
  We will assess the normal values of resting microvascular resistances using a frequentistic approach and study their associations with comorbidities and clinical parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Cardiology, Cardiology I, university hospital Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Upon legitimate request